CLINICAL TRIAL: NCT07334522
Title: Effect of Distraction Technique Using Virtual Reality on Pain and Anxiety Level During Needle Insertion in Arteriovenous Fistula Among Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Virtual Reality Distraction for Pain and Anxiety in Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karbala University (Other)
Responsible Party: Principal Investigator, Astabraq Rassoul Hussein Abass, Graduate Researcher, Ministry of Health, Iraq
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOK.CON.25.0100
Record Dates: First submitted 2026-01-01; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study will employ a randomized controlled trial using the Solomon four-group design. A total of 150 hemodialysis patients will be recruited and randomly allocated into four groups across two dialysis centers. The design includes two groups with pre-test and post-test measurements and two groups with post-test only, allowing control for pre-test sensitization and strengthening internal validity.
  The intervention protocol involves the use of virtual reality distraction as follows:
  * 2 minutes before needle insertion: patients wear the VR headset to establish immersion.
  * 3 minutes during needle insertion: VR continues throughout the cannulation procedure.
  * Immediately after completion of needle insertion: the VR headset is removed.
  Measurement Strategy
  * Anxiety: assessed using the Visual Analogue Scale for Anxiety (VAS-A), measured before and after the intervention (for pre-test groups).
  * Pain: assessed using the Visual Analogue Scale (VAS), measured only after the
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Participants in this group will receive distraction therapy using Virtual Reality (VR) glasses during the AVF insertion. The VR session starts 2 minutes before the procedure and continues for 3 minutes during the insertion. Utilizing the Solomon Four-Group Design, this group is randomly subdivided into two subgroups: in Subgroup A, anxiety is assessed before the intervention, while in Subgroup B, no pre-test assessment is performed. Both subgroups undergo post-test measurement for pain and anxiety immediately after the procedure.
  Interventions: Device: Virtual Reality
- Control Group (Active Comparator): Participants in this group will receive standard routine nursing care for AVF insertion without any additional distraction techniques. Utilizing the Solomon Four-Group Design, this group is randomly subdivided into two subgroups: in Subgroup C, anxiety is assessed before the procedure, while in Subgroup D, no pre-test assessment is performed. Both subgroups undergo post-test measurement for pain and anxiety immediately after the procedure
  Interventions: Other: standard of care

INTERVENTIONS:
Device: Virtual Reality — The intervention involves using VR glasses to provide audiovisual distraction. Participants will watch a 360-degree underwater video with calming music. The VR session starts 2 minutes before the procedure and continues for 3 minutes during the insertion
  Arms: Virtual Reality Group
Other: standard of care — Routine nursing care for AVF insertion, including skin disinfection and needle insertion according to the hospital's standard protocols, without any additional distraction techniques.
  Arms: Control Group

SUMMARY:
1. Assess pain and anxiety levels in hemodialysis patients during arteriovenous fistula needle insertion.
2. Determine the effect of the distraction technique using virtual reality on pain and anxiety levels during arteriovenous fistula needle insertion in hemodialysis patients.
3. Find out the differences in the level of pain and anxiety after using virtual reality with regard to the demographic and clinical data of the sample.

DETAILED DESCRIPTION:
Kidney Failure Requiring Replacement Therapy (KFRT) is a growing global health challenge. In 2023, the number of global cases of KFRT reached 4.59 million, affecting approximately 5 million people worldwide. Regionally, the burden is significant, with 230,000 cases reported in North Africa and the Middle East, and specifically 8,800 cases in Iraq.

Hemodialysis remains the primary life-sustaining treatment for these patients. To perform hemodialysis efficiently, a reliable vascular access is required, with the arteriovenous fistula (AVF) being the gold standard. However, the procedure requires the insertion of large-gauge needles into the fistula repeatedly (usually three times a week), which is often associated with significant pain and distress.

Needle phobia, anticipatory anxiety, and procedure-related pain are common challenges among hemodialysis patients. Unmanaged pain and anxiety can lead to poor adherence to treatment, adverse physiological responses (such as hypertension and tachycardia), and a reduced quality of life.

Virtual Reality (VR) is an immersive technology that draws the patient's attention away from the noxious stimulus by creating a simulated environment. The study aims to evaluate the efficacy of VR as a distraction method to reduce pain and anxiety during AVF cannulation in hemodialysis patients compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with End-Stage Renal Disease (ESRD) on hemodialysis.
* Patients using a functioning arteriovenous fistula (AVF).
* Conscious, oriented, and able to communicate.
* Normal or corrected vision and hearing suitable for VR use.
* Patients capable of giving written informed consent.

Exclusion Criteria:

* History of motion sickness, seizures, or epilepsy.
* Use of Central Venous Catheter (CVC) or Arteriovenous Graft (AVG).
* Use of analgesics or sedatives within 4 hours before the procedure.
* Facial wounds or eye infections preventing VR use.
* Hemodynamic instability or cognitive impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
pain intensity | Immediately after the needle insertion procedure
  Pain intensity will be assessed using the Visual Analog Scale (VAS). This scale consists of a 10-cm horizontal line where 0 represents "no pain" and 10 represents "worst possible pain." Participants will mark their perceived pain level on the line immediately after the needle insertion and removal of the VR glasses.
Anxiety Level | Immediately after the needle insertion procedure
  The anxiety level will be assessed using the Visual Analog Scale (VAS) for Anxiety. This scale consists of a 10-cm horizontal line, where 0 indicates "no anxiety" and 10 indicates "worst possible anxiety." Participants will be asked to place a mark on the line corresponding to their perceived anxiety level immediately after the needle insertion and removal of the VR glasses.

CONTACTS AND LOCATIONS:
Overall Officials: Astabraq R Hussein, MGS, Principal Investigator — kerbala heath department
Locations (2):
- Iraq (2):
  - Imam Al-Hassan Al-Mujtaba Teaching Hospital, Karbala
  - Imam Al-Hussain Teaching Hospital, Karbala

IPD SHARING:
Plan to Share IPD: No